CLINICAL TRIAL: NCT07105059
Title: Teclistamab and Mezigdomide for Relapsed/Refractory Multiple Myeloma
Brief Title: A Study of Teclistamab and Mezigdomide in People With Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-393
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
Keywords: Teclistamab; Mezigdomide; Relapsed or refractory multiple myeloma; 24-393; MATRIX (Mezigdomide And Teclistamab to Relieve Immune eXhaustion)
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Intervention Model Description: The trial will enroll a total of 18 patients, combined for the dose escalation and expansion cohorts, over a 24 month period.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Teclistamab and Mezigdomide (Experimental): The trial treatment will start with 14 days of mezigdomide priming to sensitize the myeloma cells to the bispecific antibody treatment and to stimulate and activate T-cells. After mezigdomide priming, patients will go through the step-up dosing with teclistamab- followed by combination treatment with both drugs.
  Interventions: Drug: Teclistamab; Drug: Mezigdomide

INTERVENTIONS:
Drug: Teclistamab — After the priming, patients will start Teclistamab step up dosing. Mezigdomide will not be given during the Teclistamab step up. After the priming and step-up, patients will start combination treatment with Teclistamab and Mezigdomide.
Drug: Mezigdomide — Start with 14 days of Mezigdomide. After the priming and step-up, patients will start combination treatment with Teclistamab and Mezigdomide.

SUMMARY:
The researchers are doing this study to find out whether combining teclistamab and mezigdomide is a safe and effective treatment approach in people with relapsed/refractory multiple myeloma (MM).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with relapsed or refractory multiple myeloma who have been treated with a proteasome inhibitor, an IMiD, and an anti-CD38 antibody. Patients who have been treated with at least 2 prior lines of therapy are eligible. Multiple myeloma is defined by the International Myeloma Working Group (IMWG) updated criteria.
2. Patients need to have measurable disease defined by one or more of the following:

   1. Serum myeloma (M)-protein greater than or equal to 0.5 g/dL (5 g/L).
   2. Urine M-protein greater or equal to 200 mg/24 h.
   3. Involved light chain (either kappa or lambda) >10 mg/dL with an abnormal kappa: lambda ratio
   4. Plasmacytoma(s) that is new or definitely increased verified by imaging or biopsy.

      Increase is defined as a 50% and at least 1 cm increase as measured serially by the sum of the products of the cross-diameters of the measurable lesion.
   5. A bone marrow biopsy demonstrating >30% infiltration of clonal plasma cells.
3. Patients who have received prior BCMA-directed therapy > 90 days prior including antibody drug conjugates or chimeric antigen receptor T-cell [CAR T] are eligible. BCMA presence on the cell surface should be confirmed in patients who have been treated with prior BCMA targeted therapies. Prior treatment with BCMA targeted bispecific antibodies is not allowed.
4. Patients who have received bispecific antibodies >60 days prior with targets other than BCMA are eligible.
5. Patients who have received allogeneic stem cell transplantation >6 months prior are eligible.
6. Age ≥18 years.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-1. PS-2 is permitted if PS is due solely to bone pain.
8. Fulfil the criteria for Adequate Organ System Function Based on Safety Assessments:

   Hematologic:
   * Hemoglobin ≥8 g/dL (without prior RBC transfusion within 7 days before the laboratory test; recombinant human erythropoietin use is permitted)
   * Absolute neutrophil count (ANC) ≥1.0 × 109/L (prior growth factor support is permitted but must be without support for 7 days for G-CSF or GM-CSF and for 14 days for pegylated-G-CSF) before the screening and laboratory test
   * Platelets ≥75 × 10^9/L in participants in whom <50% of bone marrow nucleated cells are plasma cells and ≥50×109 /L in participants in whom ≥50% of bone marrow nucleated cells are plasma cells (without transfusion support or thrombopoietin receptor agonist within 7 days before the screening laboratory test)

   Chemistry:
   * Total bilirubin ≤2 × ULN; except in subjects with congenital bilirubinemia, such as Gilbert syndrome (in which case if total bilirubin is >2×ULN, then direct bilirubin ≤1.5×ULN is required)
   * AST and ALT ≤2.5 × ULN
   * eGFR ≥30 mL/min Calculated by CKD-EPI formula adjusted for body surface area (BSA): (mL/min/1.73 m2) x BSA/1.73)
   * Serum calcium corrected for albumin ≤14 mg/dL (≤3.5 mmol/L) or free ionized calcium ≤6. mg/dL (≤1.6 mmol/L)
9. Resolved acute effects of any prior therapy to baseline severity or CTCAE Grade ≤ 1, with the exception of peripheral neuropathy attributable to bortezomib.
10. Female participants: A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

    ° Is not a woman of childbearing potential (WOCBP)

    Nonchildbearing potential is defined as follows (by other than medical reasons):
    * ≥45 years of age and has not had menses for >1 year
    * Patients who have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
    * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure OR
    * Is a WOCBP and agrees to use two different contraceptive methods that are highly effective (with a failure rate of <1% per year), preferably with low user dependency , during the intervention period and for at least 6 months after the last dose of study intervention.
    * WOCBP must have two negative serum or urine pregnancy tests with 10-14 days in between prior to treatment with mezigdomide. The latter must be within 15 days of starting mezigdomide. WOCBP must agree to use two highly effective methods of contraception (i.e. copper-containing intrauterine device, established use of oral, inserted, injected or implanted hormonal method of contraception, or male/female sterilization, etc.
    * WOCBP must agree not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.

    The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with a nearly undetected pregnancy. Pregnancy prevention while on mezigdomide treatment is All WOCBP must agree and adhere to all testing and contraception requirements in the mezigdomide Global Pregnancy Prevention Plan (PPP). Duration of contraception for WOCBP must be in accordance with the mezigdomide Global PPP
11. Male participants: Male participants are eligible to participate if they agree to the following: male participants must agree to practice complete abstinence or agree to use a condom during sexual contact with a pregnant partner or an WOCBP while taking mezigdomide, during dose interruptions, and for 28 days after the last dose of mezigdomide, even if they have undergone a successful vasectomy (ie, with documented azoospermia 90 days after the procedure). See mezigdomide Global PPP, Appendix 3. Male participants must agree not to donate sperm for the purpose of reproduction during this period.
12. Signed and dated Informed Consent by study participant.
13. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other procedures.

Exclusion Criteria:

1. Prior treatment with a BCMA targeted bispecific antibody
2. Prior treatment with mezigdomide
3. Systemic anti-myeloma therapy (including systemic steroids) within ≤14 days, or plasmapheresis within 7 days prior to the first dose of study drug.
4. Use of an investigational drug within 21 days or five half-lives (whichever is longer) preceding the first dose of study drug.
5. Radiation therapy within ≤14 days prior to study entry (bone lesions requiring radiation may be treated with limited [i.e., ≤ 25% of bone marrow in field] radiation therapy during this period).
6. Live, attenuated vaccine or investigational vaccine within 4 weeks before the first dose of study drug. Non-live or non-replicating vaccines authorized for emergency use (eg, COVID-19) by local health authorities are allowed
7. Patients with a history of autologous stem cell transplant within 60 days or allogeneic stem cell transplant within 6 months prior to study enrollment.
8. Patients who received CAR T therapy within 90 days prior to study enrollment
9. Patients with primary AL amyloidosis will be excluded.
10. Participant must not have had major surgery ≤4 weeks prior to initiating study treatment.
11. Evidence of active internal bleeding.
12. Presence of active renal condition. Participants with isolated proteinuria resulting from multiple myeloma are eligible, provided they fulfill criteria given
13. Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, or otherwise stable chronic liver disease per investigator's assessment).
14. Subject has active or prior history of malignancy, other than multiple myeloma, unless the subject has been free of the disease or medically stable for ≥ 2 years. The only allowed exceptions are the below listed malignancies treated within the last 24 months and that are considered cured:

    * Non-muscle invasive bladder cancer
    * Non-melanoma skin cancers treated with curative therapy or localized melanoma treated with curative surgical resection alone
    * Carcinoma in situ of the cervix
    * Carcinoma in situ of the breast
    * Localized prostate cancer (M0, N0) with a Gleason Score ≤7a, treated locally only (RP/RT/focal treatment) The participant must not be receiving active therapy, other than hormonal therapy for this disease. Presence of low risk prostate cancer per NCCN on active surveillance is permitted.
15. Evidence of cardiovascular risk including any of the following:

    * Evidence of current clinically significant untreated arrhythmias, including clinically significant ECG abnormalities including 2nd degree (Mobitz Type II) or 3rd degree atrioventricular (AV) block.
    * History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within 3 months of Screening
    * Stroke, transient ischemic attack, or seizure within 6 months prior to randomization
    * Class III or IV heart failure as defined by the New York Heart Association functional classification system.
16. Known immediate or delayed hypersensitivity reaction or idiosyncratic reaction to drugs chemically related to teclistamab or mezigdomide, or any of the components of the study treatment.
17. Pregnant or lactating individual.
18. Active infection requiring treatment.
19. Participant has known human immunodeficiency virus (HIV) infection, unless the participant can meet all of the following criteria:

    1. Established antiretroviral therapy (ART) for at least 6 months and HIV viral load <400 copies/mL, and
    2. CD4+ T-cell (CD4+) counts ≥350 cells/μL, and
    3. No history of acquired immunodeficiency s-defining opportunistic infections or other acquired immune deficiency syndrome (AIDS)-defining conditions within the last 12 months and
    4. Not receiving highly active anti-retroviral therapy, and
    5. Not receiving antiretroviral therapy that may interfere with study treatment
20. Presence of hepatitis B surface antigen (HbsAg), or hepatitis B core antibody (HbcAb at Screening or within 3 months prior to first dose of study treatment). Note: Participants with positive Hepatitis B antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis B DNA test is obtained.
21. Active Hepatitis C infection as measured by positive hepatitis C virus (HCV)-RNA testing. Subjects with a history of HCV antibody positivity must undergo HCV RNA testing. The result needs to be negative for trial eligibility.
22. Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions (including lab abnormalities) that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures.
23. Administration of strong CYP3A modulators or proton-pump inhibitors (eg, omeprazole, esomeprazole, lansoprazole, pantoprazole, rabeprazole) within 2 weeks of starting study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2028-08-08 (Estimated); Study Completion 2028-08-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Dose Limiting Toxicity Assessed by CTCAE v5.0 | 1 year

SECONDARY OUTCOMES:
Overall response rate | 2 years
  assessed using the International Myeloma Working Group (IMWG) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Malin Hultcrantz, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org